CLINICAL TRIAL: NCT03439397
Title: RCT of Ballon Technique VS Selective Ophthalmic Artery Infusion For the Retinoblastoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Jing zhang, Jing Zhang, Head of Department of Interventional Radiology, Guangzhou Women and Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GZWACMC20180112
Record Dates: First submitted 2018-01-29; First posted 2018-02-20 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Retinoblastoma; IAC; Selective Ophthalmic Artery Infusion; Ballon Technique
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ballon Technique group (Experimental): Intervention：Ballon Technique
  Interventions: Device: Ballon Technique
- SOAI group (Active Comparator): Intervention：Selective Ophthalmic Artery Infusion
  Interventions: Device: SOAI

INTERVENTIONS:
Device: Ballon Technique — Ballon Technique
  Arms: Ballon Technique group
Device: SOAI — SOAI
  Arms: SOAI group

SUMMARY:
Retinoblastoma is the most common intraocular tumor in children..IAC--Targeted Treatment for Intraocular Retinoblastoma,Is minimally invasive procedure that infuse chemotherapy select into the ophthalmic artery, its can increasing the drug concentration reaching the tumor and reducing systemic toxicity compared with traditional intravenous treatment.: one is Ballon technique , another is selective ophthalmic artery infusion.This study evaluates the difference of Ballon technique and selective ophthalmic artery infusion effect in the treatment of retinoblastoma. Half of participants will receive, Ballon technique while the other half will receive selective ophthalmic artery infusion

DETAILED DESCRIPTION:
Delivering the chemotherapeutic agent in the arterial system through the ophthalmic artery transforms the treatment of retinoblastoma from systemic chemotherapy to local chemotherapy. Two alternative means can be used,The purpose of this study is to show that Ballon technique and SOAI delivered directly through the artery supplying the eye (ophthalmic artery) to patients with retinoblastoma is a safe and effective treatment.

ELIGIBILITY:
Inclusion Criteria:

1. No age limit, no gender limit, monocular or binocular affected;
2. New diagnosed cases, without any previous treatment;
3. Clinical diagnosed as retinoblastoma, and in group C, D or E according to IIRC standard; Binocular affected with one eye enucleated;
4. Normal bone marrow function
5. Normal liver function
6. Normal kidney function
7. Normal coagulation function
8. To be willing to take part in the clinical trial and sign the informed consent form; 9. To be willing to have these tumor sites surgically removed and do the follow up accordingly.

Exclusion Criteria:

1. Diagnosis is not clear;
2. With other sever ocular diseases (for example: neovascular glaucoma, iris neovascularization);
3. With sever systemic diseases, include abnormal liver or kidney function, abnormal routine blood test or coagulation function, congenital heart diseases and dysaudia;
4. Took part in other clinical study within 3 months;
5. Refuse to take part in this clinical study;
6. Is not willing to do the follow up accordingly or follow up less than 2 times.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 496 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Globe salvage rate (Eyes saved/Eyes treated) | Three years from intervention
  Event defined as the need for external beam enucleation，To assess the saving of eyes affected with IAC for patients who would have been candidates for enucleation

SECONDARY OUTCOMES:
Visual pathway function | Three years from intervention
  Evaluation of visual pathway function will be measured composite using visual acuity, electroretinogram, visual evoked potential, and functional magnetic resonance imaging
complications | Three years from intervention
  Short and long term complications

CONTACTS AND LOCATIONS:
Overall Officials: huiming xia, Study Director — Guangzhou Women and Children's Medical Center

IPD SHARING:
Plan to Share IPD: No